CLINICAL TRIAL: NCT04442282
Title: Difficulties in Emotion-regulation and Interpersonal Problems, and Their Association With Anxiety and Depression During and After the COVID-19 Pandemic
Brief Title: Difficulties in Emotion-regulation and Interpersonal Problems During and After the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Sverre Urnes Johnson, Associate Professer Sverre Urnes Johnson, University of Oslo
Other Study IDs: REK125510 (5)
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Anxiety; Depression; Interpersonal Problem; Emotion Regulation
MeSH Terms: conditions — Anxiety Disorders; Depression; Emotional Regulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Central indicators of psychological functioning such as difficulties in emotion regulation and habitual problems in one's relating to others are likely to have been substantially impacted by the COVID-19 amelioration measures of societal lock-down and physical (ne social) distancing. In turn, as these amelioration measures have been relaxed, that impact will presumably be reduced, gradually returning these factors to pre-crisis levels. Also, these factors are likely to predict mental health outcomes such as symptoms of depression and anxiety throughout the pandemic and beyond, so that levels of emotion regulation difficulties and interpersonal problems early on will predict later symptom status. Similarly reductions in such difficulties during the various phases of the outbreak will be associated with a concurrent reduction in psychological symptoms and reduced symptom levels at later stages.

DETAILED DESCRIPTION:
Hypotheses/Research questions:

H1: There will be a significant decrease in emotion-regulation difficulties (DERS) and interpersonal problems from T1 to T2.

Exploratory: Examine the difference in interpersonal problems and DERS among different sub-groups before and after the COVID-19 pandemic

H2: Higher level at T1 and less reduction from T1 to T2 in emotion-regulation difficulties and interpersonal problems will be associated with less reduction in anxiety and depression from T1 to T2, above and beyond, demographic variables (age, gender, education).

Exploratory: Explore the different octants of IIP as predictors of changes for anxiety and depression.

This study is part of 'The Norwegian COVID-19, Mental Health and Adherence Project', involving multiple studies.

Statistical models:

Repeated surveys like the present one typically have high drop-out and substantial missing data. Therefore, we will use mixed models instead of paired t-tests, repeated measures ANOVAs, and ordinary linear regression to analyze the data. Mixed models use maximum likelihood estimation, which is the state of the art approach to handle missing data (Schafer & Graham, 2002). Especially if data are missing at random, which is likely in our survey, mixed models give more unbiased results than the other analytic methods (O'Connel et al., 2017).

In preliminary analyses, and for each of the dependent variables (GAD-7 and PHQ-9, DERS , IIP), the combination of random effects and covariance structure of residuals that gives the best fit for the "empty" model (the model without fixed predictors except the intercept) will be chosen. Akaike's Information Criterion (AIC) will used to compare the fit of different models. Models that give a reduction in AIC greater than 2 will be considered better (Burnham & Anderson, 2004). The program SPSS 25.0 will be used (IBM Corp, 2018).

First, H1 about decrease in DERS and IIP, GAD-7 and PHQ will be tested by using anxiety or depression as dependent variable in a model using time (T1 period = 0, T2 period = 1) as a predictor. Second, demographic group variables will be added as predictors. Third, the initial (T1) levels of DERS and IIP as constant covariates will be added, together with the interactions of these constant covariates with time. These interactions represent tests of H2 about the covariates predicting change in anxiety and depression. Finally, the T2 levels of DERS and IIP as constant covariates will be added, together with the interactions of these constant covariates with time. These interactions represent tests of H2 about the change in the covariates from T1 to T2 predicting change in anxiety and depression from T1 to T2s.

Transformations Depending on degree of skewness compared to theoretical possibilities and interpretations, variables will be assessed in their original and validated format as is recommended practice, as long as this is possible. As this study examines psychopathology levels amongst a general population (and not a clinical population), we do expect a skewed data. We will attempt to assess these variables in their original and validated format as is recommended practice, as long as this is possible. However, if this is not possible to the statistical assumptions behind the analyses, transformation may be needed to apply interval-based methods. Alternatively a non-parametric test will be used.

Inference criteria

Given the large sample size in this study, we pre-define our significance level:

p < 0.01 to determine significance

Missing data Maximum likelihood

Sensitivity analyses Sensitivity analyses will be conducted after selecting a random sample of participants to reflect the proportion of subgroups in the Norwegian adult population.

Exploratory:

Questions addressed in the future paper which is not pre-specified will be defined as exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all adults including those of 18 years and above,
* Who are currently living in Norway and thus experiencing identical NPIs, and
* Who provide digital consent to partake in the study.

Exclusion Criteria:

* Children and adolescents (individuals below 18)
* Adults not residing in Norway during the measurement period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: General population in Norway.
Sampling Method: Probability Sample
Enrollment: 5041 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-07-13 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Data is set to be collected starting from 22th of June. The data collection period will last no longer than three weeks depending on the response to the questionnaire
  The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) is used to measure symptoms of depression in accordance with the diagnostic criteria for major depressive disorder. The questionnaire consists of nine items where each is scored on a four-point Likert scale (0-3), with the range of scores from 0 to 27. Higher scores indicate greater depression severity, and scores above 10 are considered as the cut-off that indicating that the patient is within the depressive area.
The Generalized Anxiety Disorder - 7 | Data is set to be collected starting from 22th of June. The data collection period will last no longer than three weeks depending on the response to the questionnaire
  The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006) is a questionnaire consisting of seven items measuring symptoms of anxiety and worry. The items are scored on a four-point Likert scale (0-3), with the scores ranging from 0 to 21. Specific cut-off for Norwegian samples have been found yielding a cut-off of 8 and above for high sensitivity and specificity (Johnson, Ulvenes, Øktedalen & Hoffart, 2019).
  The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006) is a questionnaire consisting of seven items measuring symptoms of anxiety and worry. The items are scored on a four-point Likert scale (0-3), with the scores ranging from 0 to 21. Specific cut-off for Norwegian samples have been found yielding a cut-off of 8 and above for high sensitivity and specificity (Johnson, Ulvenes, Øktedalen & Hoffart, 2019).
Difficulties in Emotion Regulation Scale | Data is set to be collected starting from 22th of June. The data collection period will last no longer than three weeks depending on the response to the questionnaire
  6 items from DERS (Gratz & Roemer, 2004)
Interpersonal problems | Data is set to be collected starting from 22th of June. The data collection period will last no longer than three weeks depending on the response to the questionnaire
  17 Items from IIP-64 (Horowitz et al. 2000)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Andrè Solbakken, PhD, Principal Investigator — University of Oslo; Jon Monsen, PhD, Principal Investigator — University of Oslo; Asle Hoffart, PhD, Principal Investigator — University of Oslo & Modum Bad; Omid Ebrahimi, Mr, Principal Investigator — University of Oslo & Modum Bad

IPD SHARING:
Plan to Share IPD: No